CLINICAL TRIAL: NCT02102217
Title: PREdiction of Complications: A Step-up Approach, CRP First Followed by CT-scan Imaging to Ensure Quality Control After Major Abdominal Surgery
Brief Title: the PRECious Trial: PREdiction of Complications
Acronym: PRECious
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Amsterdam UMC, location VUmc (Other)
Responsible Party: Principal Investigator, J. Straatman, Drs. J. Straatman, Amsterdam UMC, location VUmc
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Treatment
Other Study IDs: Pro14/23
Record Dates: First submitted 2014-03-19; First posted 2014-04-02 (Estimated); Last update posted 2020-11-06 (Actual); Status verified 2020-11

CONDITIONS: Postoperative Complications
Keywords: Major Abdominal Surgery; C-reactive protein; Computed Tomography; Quality Control; Postoperative complications
MeSH Terms: conditions — Postoperative Complications

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Precious arm (Experimental): Postoperative controls according to the PRECious protocol, which entails standardized measurement of CRP levels on postoperative day three, four and five. If CRP levels exceed 140 mg/l additional CT-scan imaging will be conducted.
  Interventions: Procedure: PRECious
- Control (No Intervention): Standard postoperative controls. Additional testing will only be conducted on demand.

INTERVENTIONS:
Procedure: PRECious — Standardized measurement of serum CRP levels on postoperative day 3,4 and 5.
  Arms: Precious arm

SUMMARY:
20% of patients who undergo major abdominal surgery will have a major complication, which requires invasive treatment and is associated with increased mortality, morbidity, hospital stay and intensive care stay. A quality control algorithm after Major Abdominal Surgery (MAS) aimed at early identification of patients at risk of developing major complications can decrease associated morbidity and mortality. Literature studies show promising results for C-reactive protein as an early marker for postoperative complications, however clinical significance has yet to be determined. Here the investigators propose a randomized clinical trial in order to determine the effect of postoperative monitoring with standardized CRP measurements on postoperative morbidity and mortality, if CRP levels exceed 140 mg/L additional CT-scan imaging will be conducted.

DETAILED DESCRIPTION:
Major Abdominal Surgery (MAS) may be defined as a surgical resection performed on colorectal, hepato-pancreatico-biliary and upper-GI organs with either primary anastomosis and/or ostomy. In patients undergoing MAS postoperative complications are reported in up to 40% of patients. Around 20% of all MAS patients have a major complication, which requires invasive treatment such as reoperation, percutaneous drainage and intensive care admission. Major complications further increase morbidity and mortality after major abdominal surgery, leading to longer intensive care and hospital stay, unplanned open procedures and creation of ostomies and possible increased cancer recurrence rates and costs.

In current postoperative practice median time to clinical diagnosis of a postoperative complication is approximately eight days. A delay in diagnosis of complications increases morbidity and mortality related to major complications. Whereas early diagnosis of postoperative septic complications, before clinical deterioration, is associated with a decrease in the associated morbidity and mortality. An early detection of septic complications is challenging and may clinically and serologically, as well while using imaging techniques, be hard to distinguish from the physiological and postoperative systemic inflammatory response syndrome (SIRS). Furthermore clinical risk assessment appears to have a low predictive value for major complications such as anastomotic leak. This further stresses the need for a standardized Quality Control algorithm after MAS.

Noteworthy is that nowadays no standard Quality Control tests or protocols are available after MAS to differentiate between a normal and a complicated postoperative course.

In the search for a marker in early diagnosis of postoperative complications several biomarkers have been assessed, such as interleukin 6 (IL-6), Tumour necrosis factor α (TNF-α), procalcitonin, white blood cell count (WBC) and C-reactive protein (CRP).

WBC showed no significant differences between patients with an uncomplicated versus complicated postoperative course. WBC is therefore not useful in a standardized quality control algorithm. Procalcitonin, IL-6 and TNF-α have been assessed as markers of postoperative sepsis. However, compared to CRP they achieve similar results in predicting major complications after MAS. Moreover, taking into account the higher cost and limited availability of testing for procalcitonin, IL-6 and TNF-α levels, we further focussed on the use of CRP in a postoperative standardized quality control algorithm.

CRP is well established as a marker for infections and complications and showed promising results . It is an acute phase protein, synthesized in the liver, under stimulation of IL-6 and TNF-α in inflammatory processes, which amongst others enhances phagocytosis of bacteria by macrophages. In healthy individuals, CRP level is <1 mg/L. In mild inflammation it can rapidly reach over 40 mg/L and even over 400 mg/L have been detected in severe inflammatory response, sepsis or burns. CRP levels are also raised as a consequence of operative trauma, and it is even suggested that the level of postoperative CRP is proportional to the length of the operation, amount of operative trauma and intra-operative complications . A peak in postoperative CRP levels is observed 48-72 hours after surgery. In uneventful cases, the levels decrease after this peak. Furthermore, plasma half-life of CRP is 19 hours and is independent of diet, diurnal rhythm or organ function. Circulating CRP levels are therefore only determined by their rate of synthesis. Based on these characteristics, CRP might be a promising valuable marker for the grade of inflammation related to postoperative complications.

Several studies have assessed the use of CRP as a marker for postoperative complications after major abdominal surgery. Established cut-off CRP levels serving as markers for infective complications range from 140 mg/L to 170 mg/L on postoperative day (POD) 3. Regarding anastomotic leakage in colorectal patients, the cut-off for CRP levels have been proposed at 190 mg/L on POD 3and 125 mg/l for POD 4. Published variations in cut-offs for CRP levels are related to differing positive and negative predictive values.

The largest retrospective series included 1187 patients that had undergone colorectal surgery. They calculated a cut-off of 123 mg/L as a marker for all septic complications, yet they did not differentiate between minor and major complications. A recent meta-analysis established a cut-off of 172 mg/l on POD 3 as a marker for anastomotic leakage. Definitions regarding anastomotic leak vary widely among literature, which limits reproducibility and excludes patients that require re-intervention for other complications. Therefore our interest lies in diagnosing all major complications that require invasive treatment, as classified by grades 3-5 in the Clavien Dindo classification.

Based on our own systematic review and pooled-analysis of 1427 patients that underwent MAS, a level of 140 mg/l is proposed as cut-off for postoperative days 3,4 and 5 as a marker for major complications, with an overall sensitivity of 81,7% and a sensitivity of 61,6% Serum CRP is non-specific for location, thus additional imaging is required. Computed Tomography (CT) is the current imaging modality of choice. In our retrospective data, CT-scans showed a sensitivity of 91,7% and specificity of 100% for diagnosis of major complications, this is conformed in literature. Moreover, in the study conducted by Eckmann et al. CT-scan imaging showed a sensitivity of 97%. Another recent study established CT-scan imaging as the preferred modality in diagnosis of anastomotic leakage.

In 2008, Den Dulk et al. implemented a standardized scoring system for the clinical status of patients undergoing colorectal surgery. With this system they decreased the time between surgery and diagnosis of anastomotic leakage from 8 to 6 days, thereby decreasing mortality from 39% to 24% (p=0,24). Further supporting the role for a standardized postoperative quality control algorithm following MAS. However the search for an optimal algorithm continues.

CRP and CT scanning have shown to be able to differentiate between uncomplicated and complicated postoperative courses. Currently their use is only on demand. The here presented PRECious protocol is a postoperative Quality Control algorithm, which aims at early diagnosis and treatment of patients with major complications.

ELIGIBILITY:
Inclusion Criteria:

* Age equal to or above 18 years
* Planned elective MAS
* Written and oral informed consent

Exclusion Criteria:

* Acute MAS
* ASA classification equal to four or higher
* Insufficient Dutch language skills
* contrast allergies
* glomerular filtration rate (GFR) < 60 ml/min/1,73m2

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 525 (Actual)
Dates: Start 2015-12; Primary Completion 2020-05 (Actual); Study Completion 2020-09 (Actual)

PRIMARY OUTCOMES:
Morbidity and mortality after major complications | one year
  Combined Primary outcome, entailing both:
  1. Mortality; during 12 month follow-up
  2. Morbidity associated with major complications and after reoperation within 12 months after index operation. Including: Fistula, Wound dehiscence/incisional hernia/open abdomen, bowel obstruction or herniation, abscess, abdominal compartment syndrome, perforation of visceral organ, unplanned enterostomy, enterostomy dysfunction due to prolapse, stenosis or retraction, myocardial infarction, pulmonary embolus, respiratory insufficiency; necessitating mechanical ventilation, cerebrovascular accident, renal failure, urosepsis; urinary tract infection with positive urine and blood cultures and circulatory shock, upper GI bleeding needing intervention of any type, intra-abdominal bleeding, anastomotic leak after relaparotomy

SECONDARY OUTCOMES:
Quality of life questionnaires | 3,5 days, 3 and 12 months postoperatively
  Quality of life questionnaires will be conducted 3 and 5 days postoperatively, and during follow-up after 3 and 12 months. Questionnaires consist of the EQ-5D (EuroQol), SF-36 (Short-Form 36) and GIQLI (GastroInstestinal Quality of Life Index).
Add-on value of CRP | postoperative days 3,4 and 5
  During rounds, before CRP levels are measured, the attending physician grades patients on a scale of 1 to 10 (one being a healthy patient, ten being a patient at risk of acute death).
Length of stay | Up to one year after randomization
  total length of hospital stay in days (n)
Length of Intensive Care admission | up to one year after randomization
  total stay on the Intensive Care Unit in days (n)
Cost-efficiency | one year
  Total costs in both study arms regarding surgery, admission, additional testing, re-interventions

CONTACTS AND LOCATIONS:
Overall Officials: Jennifer Straatman, MD, Principal Investigator — VU Medisch Centrum; Donald van der Peet, MD, PhD, Principal Investigator — VU Medisch Centrum
Locations (1):
- VU Medical Center, Amsterdam, North Holland, Netherlands

REFERENCES:
- [Derived] Straatman J, Cuesta MA, Schreurs WH, Dwars BJ, Cense HA, Rijna H, Sonneveld DJ, den Boer FC, de Lange-de Klerk ES, van der Peet DL. The PRECious trial PREdiction of Complications, a step-up approach, CRP first followed by CT-scan imaging to ensure quality control after major abdominal surgery: study protocol for a stepped-wedge trial. Trials. 2015 Aug 28;16:382. doi: 10.1186/s13063-015-0903-y. PMID 26314740